CLINICAL TRIAL: NCT06798558
Title: Phase II Study of Neoadjuvant Lu-177-PSMA-617 in Patients With High Risk Localized Prostate Cancer Undergoing Radical Prostatectomy
Brief Title: Neoadjuvant Lu-177-PSMA-617 in Patients With High Risk Localized Prostate Cancer Undergoing Radical Prostatectomy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Lombardi Comprehensive Cancer Center (Other); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRELUDE; CAAA617A1US07T (Other Grant/Funding Number: Novartis); Pro2024-0079 (Other: HMH)
Record Dates: First submitted 2025-01-17; First posted 2025-01-29 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Prostate Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lu-177-PSMA-617 Treatment (Experimental): Patients will receive 2 cycles of Lu-177-PSMA-617 (PluvictoⓇ) administered at the dose of 7.4 GBq (±10%), once every 6 weeks (±1 week)
  Interventions: Drug: Lu-17-PSMA-617

INTERVENTIONS:
Drug: Lu-17-PSMA-617 — Lu-17-PSMA-617 administration

SUMMARY:
Male adults with a confirmed diagnosis of prostate adenocarcinoma who meet criteria for localized high risk prostate cancer according to the NCCN guidelines and who are eligible for prostatectomy will be invited to participate. Criteria for high-risk prostate cancer include patients with preoperative prostate biopsy score of Gleason 8 (GS8) (Grade group 4 [GG4]) or higher. Patients also need to have a positive PSMA scan on 68-Ga-PSMA-11 PET/CT scan.

DETAILED DESCRIPTION:
The PRELUDE trial is a prospective, non-randomized, single-arm, phase 2 interventional study to assess the oncological outcomes after 2 cycles of Lu-177-PSMA-617 (PluvictoⓇ) administered at 6-week intervals before prostatectomy in patients with high risk localized prostate cancer.

Patients who meet all the inclusion criteria for the study will be enrolled to receive 2 cycles of Lu-177-PSMA-617 (PluvictoⓇ) administered at the dose of 7.4 GBq (±10%), once every 6 weeks (±1 week). Six weeks after the second cycle of Lu-177-PSMA-617 (PluvictoⓇ), patients will be eligible for radical prostatectomy with pelvic lymph node dissection and remain eligible for surgery up until 30 days from this timepoint.

Following treatment with Lu-177-PSMA-617 (PluvictoⓇ) and surgery, all participants will be followed for safety at week 3, 6, 9, 11, and 12 as well as a 30-day safety follow-up visit (FUP) and longer term safety follow-up assessments every 3 months for a period of approximately 2 years. Patients who experience disease progression will be managed according to standard treatment guidelines recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 or older.
* Patients with histologically confirmed adenocarcinoma of the prostate.
* Patients with high-risk disease defined as a preoperative prostate biopsy of Gleason Score 8 (GS8) (Grade group 4 [GG4]) or higher. Men with evidence of lymph node involvement at or below the bifurcation of the common iliac arteries (cN1) on PET-CT 68Ga-PSMA-11 are eligible.
* Pre-operative, pre-treatment PSMA scan with high expression in prostate confirmed by PET/CT 68Ga-PSMA-11 (greater than liver). Patients must not have any other PET FDG-positive sites outside the prostate.
* Patients who are able and willing to undergo surgery.
* Patients with a life expectancy of greater than 10 years. Life expectancy can be estimated using any 1 of the following tools:

  * The Social Security Administration tables:

https://www.ssa.gov/OACT/STATS/table4c6.html

* The WHO's Life Tables by country:

https://apps.who.int/gho/data/view.main.60000?lang=en

* The Memorial Sloan Kettering Male Life Expectancy tool:

https://www.mskcc.org/nomograms/prostate

* If using a life expectancy table, life expectancy should be adjusted using the clinician's assessment of overall health as follows: best quartile of health - add 50%; worst quartile of health - subtract 50%; and middle two quartiles of health - no adjustment. See the NCCN Prostate Cancer Guidelines for more information.

  * Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
  * Patients who agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agree to refrain from donating sperm, as defined below:
* With a female partner of childbearing potential who is not pregnant, men who are not surgically sterile must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for 14 weeks after the final dose of study treatment. Men must refrain from donating sperm during this same period.
* With a pregnant female partner, men must remain abstinent or use a condom during the treatment period and for 14 weeks after the final dose of study treatment to avoid potential exposure to the embryo.
* The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not adequate methods of contraception.

  * Patients who are able to comply with follow-up visits and treatment plans.
  * Patients who are able to give informed consent.

Exclusion Criteria:

* Patients with a prior history of prostate cancer treatment.
* Patients with previous treatment with PSMA-targeted radioligand therapy or any of the following within 6 months of enrollment confirmation: Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223 or hemi-body irradiation.
* Patients with distant disease (outside of local lymph nodes).
* Significant bone marrow impairment defined by leukocytes <3,000/mcL, absolute neutrophil count (ANC) <1,500/mcL, and platelet count lower than 70,000/mcL.
* Significant liver function impairment defined by total bilirubin higher than 1.5 times the upper limit of normal (ULN), andASL/ALT higher than 3 times the ULN.
* Impaired kidney function defined by glomerular filtration rate (GFR) lower than 40 mL/min, or concomitant use of nephrotoxic drugs. Kidney function based on eGFR by Modification of Diet in Renal Disease (MDRD) equation:

  * Normal renal function: participants with eGFR 90 mL/min
  * Moderate renal impairment: participants with eGFR 30 to 59 mL/min
  * Severe renal impairment: participants with eGFR 15 to 29 mL/min
* Patients with significant comorbidities that would make them poor candidates for surgery.
* Patients with evidence of metastatic disease (enlarged lymph nodes, distant metastatic sites, visceral or bone metastases, etc.).
* Patients with a history of radiation or hormone therapy to the prostate.
* Patients with a history of bleeding disorders or who are taking anticoagulant therapy.
* Patients with active infections or other contraindications for surgery.
* Patients who are unable or unwilling to give informed consent.
* Patients who are unable to comply with follow-up visits and treatment plans

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 54 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Prostate cancer down-staging following treatment with Lu-177-PSMA-617 (PluvictoⓇ) defined by Gleason Grade Group | Patients will undergo a PSMA PET/CT scans up to week 11 +/- 30 days prior to radical prostatectomy with pelvic lymph node dissection.
  Staging of prostate cancer is based on the correlation to Gleason Grade Group (GG) according to the American Joint Committee on Cancer (AJCC; 8TH edition, 2017) staging system for prostate cancer (see Appendix A). Prostate cancer downstaging is defined as the post-treatment stage less than the pre-treatment stage. Different downstaging thresholds will be applied including:
  * Complete downstaging (CD) is defined as no visible tumor in surgical sample;
  * Good response (GR) is defined as downstaging from high risk disease (GG4 or greater) to intermediate risk pathologic disease (GG2 or GG3 disease); and
  * Very good response (VGR) is defined as downstaging from high-risk disease (GG4 or greater) to low risk pathologic disease (GG1 disease).

SECONDARY OUTCOMES:
Prostate cancer down-staging following treatment with Lu-177-PSMA-617 (PluvictoⓇ) as defined by margin status, T staging, and seminal vesicle involvement | Patients will undergo a PSMA PET/CT scans up to week 11 +/- 30 days prior to radical prostatectomy with pelvic lymph node dissection.
  Staging of prostate cancer is based on the American Joint Committee on Cancer (AJCC; 8TH edition, 2017) combining the TNM staging system for prostate cancer with the Gleason Grade Group (GG)
Decrease in PSMA-avid tumor load | Patients will undergo a SOC PSMA PET/CT scans up to week 11 +/- 30 days prior to radical prostatectomy with pelvic lymph node dissection.
  Decrease in PSMA-avid tumor load is measured by comparing the extent of PSMA-avid tumor before and after Lu-177-PSMA-617 (PluvictoⓇ). High PSMA-avidity is defined as more than 2 times the liver activity. Low PSMA-avidity is defined as less than 2 times liver activity. The volumes of PSMA-avid disease will be summed up to quantify the extent of PSMA-avid tumor load before and after Lu-177-PSMA-617 (PluvictoⓇ). PSMA-positive disease is measured using 68Ga-PSMA-11 PET/CT scan.
Safety of radical prostatectomy assessed by surgical delay time | Patients will be assessed for toxicity throughout treatment with Lu-177-PSMA-617 (PluvictoⓇ) and during surgery. Following treatment with Lu-177-PSMA-617 (PluvictoⓇ) and surgery, all participants will be followed for safety with a 30-day safety follow-up
  The safety of radical prostatectomy and pelvic lymph node dissection following Lu-177-PSMA-617 (PluvictoⓇ) is defined as the surgical delay time. Surgical delay time is defined as days between the last dose of Lu-177-PSMA-617 (PluvictoⓇ) and the date of radical prostatectomy. All surgeries will be assessed by each surgeon at the end of the procedure and graded as similar to, more difficult than, or significantly more difficult than expected for a high-risk radical prostatectomy (Eapen 2023). Adverse events (AEs) of Lu-177-PSMA-617 (PluvictoⓇ) and surgery will be assessed and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 or severity grade when CTCAE grading does not exist.
Safety of radical prostatectomy assessed by rate of intraoperative and postoperative complications | Patients will be assessed for toxicity throughout treatment with Lu-177-PSMA-617 (PluvictoⓇ) and during surgery. Following treatment with Lu-177-PSMA-617 (PluvictoⓇ) and surgery, all participants will be followed for safety with a 30-day safety follow-up
  The safety of radical prostatectomy and pelvic lymph node dissection following Lu-177-PSMA-617 (PluvictoⓇ) is defined as the rate of intraoperative and postoperative complications. All surgeries will be assessed by each surgeon at the end of the procedure and graded as similar to, more difficult than, or significantly more difficult than expected for a high-risk radical prostatectomy (Eapen 2023). Adverse events (AEs) of Lu-177-PSMA-617 (PluvictoⓇ) and surgery will be assessed and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 or severity grade when CTCAE grading does not exist.
Safety of radical prostatectomy assessed by the amount of blood loss | Patients will be assessed for toxicity throughout treatment with Lu-177-PSMA-617 (PluvictoⓇ) and during surgery. Following treatment with Lu-177-PSMA-617 (PluvictoⓇ) and surgery, all participants will be followed for safety with a 30-day safety follow-up
  The safety of radical prostatectomy and pelvic lymph node dissection following Lu-177-PSMA-617 (PluvictoⓇ) is defined as the amount of blood loss. All surgeries will be assessed by each surgeon at the end of the procedure and graded as similar to, more difficult than, or significantly more difficult than expected for a high-risk radical prostatectomy (Eapen 2023). Adverse events (AEs) of Lu-177-PSMA-617 (PluvictoⓇ) and surgery will be assessed and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 or severity grade when CTCAE grading does not exist.
Safety of radical prostatectomy assessed by percentage of periprostatic adhesion | Patients will be assessed for toxicity throughout treatment with Lu-177-PSMA-617 (PluvictoⓇ) and during surgery. Following treatment with Lu-177-PSMA-617 (PluvictoⓇ) and surgery, all participants will be followed for safety with a 30-day safety follow-up
  The safety of radical prostatectomy and pelvic lymph node dissection following Lu-177-PSMA-617 (PluvictoⓇ) is defined as the percentage of periprostatic adhesion. All surgeries will be assessed by each surgeon at the end of the procedure and graded as similar to, more difficult than, or significantly more difficult than expected for a high-risk radical prostatectomy (Eapen 2023). Adverse events (AEs) of Lu-177-PSMA-617 (PluvictoⓇ) and surgery will be assessed and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 or severity grade when CTCAE grading does not exist.
Safety of radical prostatectomy assessed by the surgical length of time | Patients will be assessed for toxicity throughout treatment with Lu-177-PSMA-617 (PluvictoⓇ) and during surgery. Following treatment with Lu-177-PSMA-617 (PluvictoⓇ) and surgery, all participants will be followed for safety with a 30-day safety follow-up
  The safety of radical prostatectomy and pelvic lymph node dissection following Lu-177-PSMA-617 (PluvictoⓇ) is defined as the surgical length of time. All surgeries will be assessed by each surgeon at the end of the procedure and graded as similar to, more difficult than, or significantly more difficult than expected for a high-risk radical prostatectomy (Eapen 2023). Adverse events (AEs) of Lu-177-PSMA-617 (PluvictoⓇ) and surgery will be assessed and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 or severity grade when CTCAE grading does not exist.
Quality-of-life and sexual function changes | The EPIC-26 questionnaire will be completed by patients up to 24 months after prostatectomy
  Quality-of-life and sexual function changes following treatment with Lu-177-PSMA-617 (PluvictoⓇ) and prostatectomy will be measured using the Expanded Prostate Index Composite (EPIC)-26 questionnaire.
Biochemical recurrence of prostate cancer at 2 years | PSA levels will be measured up to 24 months after prostatectomy
  Biochemical recurrence is defined as a serum prostate-specific antigen (PSA) level more than 0.2 ng/mL on 2 consecutive measurements performed at least 3 months apart.
  Timeframe: PSA levels will be measured at screening/baseline, at the initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Yerram, MD, Principal Investigator — Hackensack Meridian Health
Locations (3):
- United States (3):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aalberts M, Stout TA, Stoorvogel W. Prostasomes: extracellular vesicles from the prostate. Reproduction. 2013 Nov 16;147(1):R1-14. doi: 10.1530/REP-13-0358. Print 2014 Jan. PMID 24149515
- [Background] Powell IJ, Dyson G, Land S, Ruterbusch J, Bock CH, Lenk S, Herawi M, Everson R, Giroux CN, Schwartz AG, Bollig-Fischer A. Genes associated with prostate cancer are differentially expressed in African American and European American men. Cancer Epidemiol Biomarkers Prev. 2013 May;22(5):891-7. doi: 10.1158/1055-9965.EPI-12-1238. Epub 2013 Mar 20. PMID 23515145
- [Background] Attard G, Murphy L, Clarke NW, Cross W, Jones RJ, Parker CC, Gillessen S, Cook A, Brawley C, Amos CL, Atako N, Pugh C, Buckner M, Chowdhury S, Malik Z, Russell JM, Gilson C, Rush H, Bowen J, Lydon A, Pedley I, O'Sullivan JM, Birtle A, Gale J, Srihari N, Thomas C, Tanguay J, Wagstaff J, Das P, Gray E, Alzoueb M, Parikh O, Robinson A, Syndikus I, Wylie J, Zarkar A, Thalmann G, de Bono JS, Dearnaley DP, Mason MD, Gilbert D, Langley RE, Millman R, Matheson D, Sydes MR, Brown LC, Parmar MKB, James ND; Systemic Therapy in Advancing or Metastatic Prostate cancer: Evaluation of Drug Efficacy (STAMPEDE) investigators. Abiraterone acetate and prednisolone with or without enzalutamide for high-risk non-metastatic prostate cancer: a meta-analysis of primary results from two randomised controlled phase 3 trials of the STAMPEDE platform protocol. Lancet. 2022 Jan 29;399(10323):447-460. doi: 10.1016/S0140-6736(21)02437-5. Epub 2021 Dec 23. PMID 34953525
- [Background] Bebelman MP, Janssen E, Pegtel DM, Crudden C. The forces driving cancer extracellular vesicle secretion. Neoplasia. 2021 Jan;23(1):149-157. doi: 10.1016/j.neo.2020.11.011. Epub 2020 Dec 14. PMID 33321449
- [Background] Becker A, Thakur BK, Weiss JM, Kim HS, Peinado H, Lyden D. Extracellular Vesicles in Cancer: Cell-to-Cell Mediators of Metastasis. Cancer Cell. 2016 Dec 12;30(6):836-848. doi: 10.1016/j.ccell.2016.10.009. PMID 27960084
- [Background] Carlsson L, Pahlson C, Bergquist M, Ronquist G, Stridsberg M. Antibacterial activity of human prostasomes. Prostate. 2000 Sep 1;44(4):279-86. doi: 10.1002/1097-0045(20000901)44:43.0.co;2-2. PMID 10951492
- [Background] Cooperberg MR, Cowan J, Broering JM, Carroll PR. High-risk prostate cancer in the United States, 1990-2007. World J Urol. 2008 Jun;26(3):211-8. doi: 10.1007/s00345-008-0250-7. Epub 2008 Mar 28. PMID 18369637
- [Background] D'Amico AV, Whittington R, Malkowicz SB, Fondurulia J, Chen MH, Kaplan I, Beard CJ, Tomaszewski JE, Renshaw AA, Wein A, Coleman CN. Pretreatment nomogram for prostate-specific antigen recurrence after radical prostatectomy or external-beam radiation therapy for clinically localized prostate cancer. J Clin Oncol. 1999 Jan;17(1):168-72. doi: 10.1200/JCO.1999.17.1.168. PMID 10458230
- [Background] D'Amico AV, Whittington R, Malkowicz SB, Fondurulia J, Chen MH, Tomaszewski JE, Wein A. The combination of preoperative prostate specific antigen and postoperative pathological findings to predict prostate specific antigen outcome in clinically localized prostate cancer. J Urol. 1998 Dec;160(6 Pt 1):2096-101. doi: 10.1097/00005392-199812010-00041. PMID 9817331
- [Background] D'Amico AV, Whittington R, Malkowicz SB, Schultz D, Blank K, Broderick GA, Tomaszewski JE, Renshaw AA, Kaplan I, Beard CJ, Wein A. Biochemical outcome after radical prostatectomy, external beam radiation therapy, or interstitial radiation therapy for clinically localized prostate cancer. JAMA. 1998 Sep 16;280(11):969-74. doi: 10.1001/jama.280.11.969. PMID 9749478
- [Background] Eapen RS, Buteau JP, Jackson P, Mitchell C, Oon SF, Alghazo O, McIntosh L, Dhiantravan N, Scalzo MJ, O'Brien J, Sandhu S, Azad AA, Williams SG, Sharma G, Haskali MB, Bressel M, Chen K, Jenjitranant P, McVey A, Moon D, Lawrentschuk N, Neeson PJ, Murphy DG, Hofman MS. Administering [177Lu]Lu-PSMA-617 Prior to Radical Prostatectomy in Men with High-risk Localised Prostate Cancer (LuTectomy): A Single-centre, Single-arm, Phase 1/2 Study. Eur Urol. 2024 Mar;85(3):217-226. doi: 10.1016/j.eururo.2023.08.026. Epub 2023 Oct 26. PMID 37891072
- [Background] Fabiani R, Johansson L, Lundkvist O, Ronquist G. Enhanced recruitment of motile spermatozoa by prostasome inclusion in swim-up medium. Hum Reprod. 1994 Aug;9(8):1485-9. doi: 10.1093/oxfordjournals.humrep.a138735. PMID 7989510
- [Background] Gafita A, Djaileb L, Rauscher I, Fendler WP, Hadaschik B, Rowe SP, Herrmann K, Calais J, Rettig M, Eiber M, Weber M, Benz MR, Farolfi A. Response Evaluation Criteria in PSMA PET/CT (RECIP 1.0) in Metastatic Castration-resistant Prostate Cancer. Radiology. 2023 Jul;308(1):e222148. doi: 10.1148/radiol.222148. PMID 37432081
- [Background] Gafita A, Rauscher I, Weber M, Hadaschik B, Wang H, Armstrong WR, Tauber R, Grogan TR, Czernin J, Rettig MB, Herrmann K, Calais J, Weber WA, Benz MR, Fendler WP, Eiber M. Novel Framework for Treatment Response Evaluation Using PSMA PET/CT in Patients with Metastatic Castration-Resistant Prostate Cancer (RECIP 1.0): An International Multicenter Study. J Nucl Med. 2022 Nov;63(11):1651-1658. doi: 10.2967/jnumed.121.263072. Epub 2022 Apr 14. PMID 35422442
- [Background] Ginini L, Billan S, Fridman E, Gil Z. Insight into Extracellular Vesicle-Cell Communication: From Cell Recognition to Intracellular Fate. Cells. 2022 Apr 19;11(9):1375. doi: 10.3390/cells11091375. PMID 35563681
- [Background] Ham WS, Chalfin HJ, Feng Z, Trock BJ, Epstein JI, Cheung C, Humphreys E, Partin AW, Han M. New Prostate Cancer Grading System Predicts Long-term Survival Following Surgery for Gleason Score 8-10 Prostate Cancer. Eur Urol. 2017 Jun;71(6):907-912. doi: 10.1016/j.eururo.2016.11.006. Epub 2016 Nov 19. PMID 27876305
- [Background] Jackson W, Hamstra DA, Johnson S, Zhou J, Foster B, Foster C, Li D, Song Y, Palapattu GS, Kunju LP, Mehra R, Feng FY. Gleason pattern 5 is the strongest pathologic predictor of recurrence, metastasis, and prostate cancer-specific death in patients receiving salvage radiation therapy following radical prostatectomy. Cancer. 2013 Sep 15;119(18):3287-94. doi: 10.1002/cncr.28215. Epub 2013 Jul 2. PMID 23821578
- [Background] Kalluri R, LeBleu VS. The biology, function, and biomedical applications of exosomes. Science. 2020 Feb 7;367(6478):eaau6977. doi: 10.1126/science.aau6977. PMID 32029601
- [Background] Kumar S, Shelley M, Harrison C, Coles B, Wilt TJ, Mason MD. Neo-adjuvant and adjuvant hormone therapy for localised and locally advanced prostate cancer. Cochrane Database Syst Rev. 2006 Oct 18;2006(4):CD006019. doi: 10.1002/14651858.CD006019.pub2. PMID 17054269
- [Background] Loeb S, Schaeffer EM, Trock BJ, Epstein JI, Humphreys EB, Walsh PC. What are the outcomes of radical prostatectomy for high-risk prostate cancer? Urology. 2010 Sep;76(3):710-4. doi: 10.1016/j.urology.2009.09.014. Epub 2009 Nov 22. PMID 19931898
- [Background] Manouchehri Doulabi E, Fredolini C, Gallini R, Lof L, Shen Q, Ikebuchi R, Dubois L, Azimi A, Loudig O, Gabrielsson S, Landegren U, Larsson A, Bergquist J, Kamali-Moghaddam M. Surface protein profiling of prostate-derived extracellular vesicles by mass spectrometry and proximity assays. Commun Biol. 2022 Dec 22;5(1):1402. doi: 10.1038/s42003-022-04349-x. PMID 36550367
- [Background] Minelli A, Ronquist G, Carlsson L, Mearini E, Nilsson O, Larsson A. Antiprostasome antibody titres in benign and malignant prostate disease. Anticancer Res. 2005 Nov-Dec;25(6C):4399-402. PMID 16334115
- [Background] Mitchell MI, Ben-Dov IZ, Liu C, Ye K, Chow K, Kramer Y, Gangadharan A, Park S, Fitzgerald S, Ramnauth A, Perlin DS, Donato M, Bhoy E, Manouchehri Doulabi E, Poulos M, Kamali-Moghaddam M, Loudig O. Extracellular Vesicle Capture by AnTibody of CHoice and Enzymatic Release (EV-CATCHER): A customizable purification assay designed for small-RNA biomarker identification and evaluation of circulating small-EVs. J Extracell Vesicles. 2021 Jun;10(8):e12110. doi: 10.1002/jev2.12110. Epub 2021 Jun 3. PMID 34122779
- [Background] Mitchell JA, Cooperberg MR, Elkin EP, Lubeck DP, Mehta SS, Kane CJ, Carroll PR. Ability of 2 pretreatment risk assessment methods to predict prostate cancer recurrence after radical prostatectomy: data from CaPSURE. J Urol. 2005 Apr;173(4):1126-31. doi: 10.1097/01.ju.0000155535.25971.de. PMID 15758720
- [Background] Schaeffer EM, Srinivas S, Adra N, An Y, Barocas D, Bitting R, Bryce A, Chapin B, Cheng HH, D'Amico AV, Desai N, Dorff T, Eastham JA, Farrington TA, Gao X, Gupta S, Guzzo T, Ippolito JE, Kuettel MR, Lang JM, Lotan T, McKay RR, Morgan T, Netto G, Pow-Sang JM, Reiter R, Roach M, Robin T, Rosenfeld S, Shabsigh A, Spratt D, Teply BA, Tward J, Valicenti R, Wong JK, Berardi RA, Shead DA, Freedman-Cass DA. NCCN Guidelines(R) Insights: Prostate Cancer, Version 1.2023. J Natl Compr Canc Netw. 2022 Dec;20(12):1288-1298. doi: 10.6004/jnccn.2022.0063. PMID 36509074
- [Background] Narang AK, Gergis C, Robertson SP, He P, Ram AN, McNutt TR, Griffith E, DeWeese TA, Honig S, Singh H, Song DY, Tran PT, DeWeese TL. Very High-Risk Localized Prostate Cancer: Outcomes Following Definitive Radiation. Int J Radiat Oncol Biol Phys. 2016 Feb 1;94(2):254-62. doi: 10.1016/j.ijrobp.2015.10.056. Epub 2015 Oct 31. PMID 26853334
- [Background] Pluvicto (lutetium lu 177 vipivotide tetraxetan) [prescribing information]. Millburn, NJ: Advanced Accelerator Applications USA Inc; October 2022.
- [Background] Pluvicto (lutetium lu 177 vipivotide tetraxetan) [product monograph]. Millburn, NJ: Advanced Accelerator Applications USA Inc; August 2022.
- [Background] Poliakov A, Spilman M, Dokland T, Amling CL, Mobley JA. Structural heterogeneity and protein composition of exosome-like vesicles (prostasomes) in human semen. Prostate. 2009 Feb 1;69(2):159-67. doi: 10.1002/pros.20860. PMID 18819103
- [Background] Ronquist G, Nilsson BO. The Janus-faced nature of prostasomes: their pluripotency favours the normal reproductive process and malignant prostate growth. Prostate Cancer Prostatic Dis. 2004;7(1):21-31. doi: 10.1038/sj.pcan.4500684. PMID 14999234
- [Background] Saez F, Motta C, Boucher D, Grizard G. Antioxidant capacity of prostasomes in human semen. Mol Hum Reprod. 1998 Jul;4(7):667-72. doi: 10.1093/molehr/4.7.667. PMID 9701789
- [Background] Sartor O, de Bono J, Chi KN, Fizazi K, Herrmann K, Rahbar K, Tagawa ST, Nordquist LT, Vaishampayan N, El-Haddad G, Park CH, Beer TM, Armour A, Perez-Contreras WJ, DeSilvio M, Kpamegan E, Gericke G, Messmann RA, Morris MJ, Krause BJ; VISION Investigators. Lutetium-177-PSMA-617 for Metastatic Castration-Resistant Prostate Cancer. N Engl J Med. 2021 Sep 16;385(12):1091-1103. doi: 10.1056/NEJMoa2107322. Epub 2021 Jun 23. PMID 34161051
- [Background] Schulman CC, Debruyne FM, Forster G, Selvaggi FP, Zlotta AR, Witjes WP. 4-Year follow-up results of a European prospective randomized study on neoadjuvant hormonal therapy prior to radical prostatectomy in T2-3N0M0 prostate cancer. European Study Group on Neoadjuvant Treatment of Prostate Cancer. Eur Urol. 2000 Dec;38(6):706-13. doi: 10.1159/000020366. PMID 11111188
- [Background] Skibinski G, Kelly RW, Harkiss D, James K. Immunosuppression by human seminal plasma--extracellular organelles (prostasomes) modulate activity of phagocytic cells. Am J Reprod Immunol. 1992 Sep;28(2):97-103. doi: 10.1111/j.1600-0897.1992.tb00767.x. PMID 1337434
- [Background] Spahn M, Joniau S, Gontero P, Fieuws S, Marchioro G, Tombal B, Kneitz B, Hsu CY, Van Der Eeckt K, Bader P, Frohneberg D, Tizzani A, Van Poppel H. Outcome predictors of radical prostatectomy in patients with prostate-specific antigen greater than 20 ng/ml: a European multi-institutional study of 712 patients. Eur Urol. 2010 Jul;58(1):1-7; discussion 10-1. doi: 10.1016/j.eururo.2010.03.001. Epub 2010 Mar 17. PMID 20299147
- [Background] Sundi D, Tosoian JJ, Nyame YA, Alam R, Achim M, Reichard CA, Li J, Wilkins L, Schwen Z, Han M, Davis JW, Klein EA, Schaeffer EM, Stephenson AJ, Ross AE, Chapin BF. Outcomes of very high-risk prostate cancer after radical prostatectomy: Validation study from 3 centers. Cancer. 2019 Feb 1;125(3):391-397. doi: 10.1002/cncr.31833. Epub 2018 Nov 13. PMID 30423193
- [Background] Sundi D, Wang VM, Pierorazio PM, Han M, Bivalacqua TJ, Ball MW, Antonarakis ES, Partin AW, Schaeffer EM, Ross AE. Very-high-risk localized prostate cancer: definition and outcomes. Prostate Cancer Prostatic Dis. 2014 Mar;17(1):57-63. doi: 10.1038/pcan.2013.46. Epub 2013 Nov 5. PMID 24189998
- [Background] Tan M, Xiong X. Continuous and group sequential conditional probability ratio tests for phase II clinical trials. Stat Med. 1996 Oct 15;15(19):2037-51. doi: 10.1002/(SICI)1097-0258(19961015)15:193.0.CO;2-Z. PMID 8896138
- [Background] Tan MT, Xiong X. A flexible multi-stage design for phase II oncology trials. Pharm Stat. 2011 Jul-Aug;10(4):369-73. doi: 10.1002/pst.478. Epub 2010 Dec 8. PMID 22328328
- [Background] Tavoosidana G, Ronquist G, Darmanis S, Yan J, Carlsson L, Wu D, Conze T, Ek P, Semjonow A, Eltze E, Larsson A, Landegren UD, Kamali-Moghaddam M. Multiple recognition assay reveals prostasomes as promising plasma biomarkers for prostate cancer. Proc Natl Acad Sci U S A. 2011 May 24;108(21):8809-14. doi: 10.1073/pnas.1019330108. Epub 2011 May 9. PMID 21555566
- [Background] Vickram S, Rohini K, Anbarasu K, Dey N, Jeyanthi P, Thanigaivel S, Issac PK, Arockiaraj J. Semenogelin, a coagulum macromolecule monitoring factor involved in the first step of fertilization: A prospective review. Int J Biol Macromol. 2022 Jun 1;209(Pt A):951-962. doi: 10.1016/j.ijbiomac.2022.04.079. Epub 2022 Apr 18. PMID 35447263
- [Background] Yang C, Guo WB, Zhang WS, Bian J, Yang JK, Zhou QZ, Chen MK, Peng W, Qi T, Wang CY, Liu CD. Comprehensive proteomics analysis of exosomes derived from human seminal plasma. Andrology. 2017 Sep;5(5):1007-1015. doi: 10.1111/andr.12412. PMID 28914500
- [Background] Yu W, Hurley J, Roberts D, Chakrabortty SK, Enderle D, Noerholm M, Breakefield XO, Skog JK. Exosome-based liquid biopsies in cancer: opportunities and challenges. Ann Oncol. 2021 Apr;32(4):466-477. doi: 10.1016/j.annonc.2021.01.074. Epub 2021 Feb 4. PMID 33548389
- [Background] Zagars GK, Pollack A, von Eschenbach AC. Prognostic factors for clinically localized prostate carcinoma: analysis of 938 patients irradiated in the prostate specific antigen era. Cancer. 1997 Apr 1;79(7):1370-80. PMID 9083160